CLINICAL TRIAL: NCT03686852
Title: Effect of Recombinant FSH Dosing Following Cori-follitropin Alfa in Patients Undergoing in Vitro Fertilization/Intra-citoplasmatic Sperm Injection: a Randomized Controlled Dose-finding Study.
Brief Title: Effect of Recombinant Follicular Stimulating Hormone (FSH) Dosing Following Cori-follitropin Alfa
Acronym: TBC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: AZ Jan Palfijn Gent (Other); Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rFSHdosingfinding.2018
Record Dates: First submitted 2018-09-25; First posted 2018-09-27 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2018-09

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group A (Active Comparator): The main difference between the groups is due to the different dose of r-FSH which will be given to pa-tients after the 7 days of CFA; namely that patients who need additional r-FSH following corifollitropin-alfa will be randomized on day 8 of the stimulation into 3 study groups. In group A, B and C, ovarian stimula-tion with Corifollitropin alfa (Elonva®, MSD) will be used for ovarian stimulation, followed by 50IU (Group A).
  Interventions: Other: same medications but different dosages
- groppo B (Active Comparator): The main difference between the groups is due to the different dose of r-FSH which will be given to pa-tients after the 7 days of CFA; namely that patients who need additional r-FSH following corifollitropin-alfa will be randomized on day 8 of the stimulation into 3 study groups. In group A, B and C, ovarian stimula-tion with Corifollitropin alfa (Elonva®, MSD) will be used for ovarian stimulation, followed by 150IU (Group B)
  Interventions: Other: same medications but different dosages
- Group C (Active Comparator): The main difference between the groups is due to the different dose of r-FSH which will be given to pa-tients after the 7 days of CFA; namely that patients who need additional r-FSH following corifollitropin-alfa will be randomized on day 8 of the stimulation into 3 study groups. In group A, B and C, ovarian stimula-tion with Corifollitropin alfa (Elonva®, MSD) will be used for ovarian stimulation, followed by 250IU (Group C) of recFSH (Puregon®, MSD).
  Interventions: Other: same medications but different dosages

INTERVENTIONS:
Other: same medications but different dosages — The main difference between the groups is due to the different dose of r-FSH which will be given to pa-tients after the 7 days of CFA; namely that patients who need additional r-FSH following corifollitropin-alfa will be randomized on day 8 of the stimulation into 3 study groups. In group A, B and C, ovarian stimula-tion with Corifollitropin alfa (Elonva®, MSD) will be used for ovarian stimulation, followed by 50IU (Group A), 150IU (Group B) or 250IU (Group C) of recFSH (Puregon®, MSD)

SUMMARY:
In the trial, women planned to be treated with 150μg corifollitropin alfa followed by rFSH in a fixed GnRH antagonist protocol will be asked to participate and sign the ICF. Corifollitropin alpha treatment will be initiated at D2-D3 of the cycle. Patients who need additional r-FSH following corifollitropin-alfa will be randomized on day 8 of the stimulation into 3 study groups. In group A, B and C, ovarian stimulation with Corifollitropin alfa (Elonva®, MSD) will be used for ovarian stimulation, followed by 50IU (Group A), 150IU (Group B) or 250IU (Group C) of recFSH (Puregon®, MSD).

DETAILED DESCRIPTION:
On day 2 or on day 3 of the cycle, blood sampling for estradiol (E2), progesterone (P), follicle stimulating hormone (FSH), luteinising hormone (LH) and human chorionic gonadotropin (hCG) levels, will be per-formed prior to the administration of corifollitropin alfa.

All the blood samples taken during the stimulation for the hormonal profile, starting from day 2, will be performed in a double tube, one for a central assessment and one for the local assessment in order to be used during the monitoring of the cycle. AMH will also be assess on day 2 of the stimulation with a blood sample that will be sent for central assessment.

Administration of the GnRH antagonist ganirelix (Orgalutran®, MSD) will be initiated on day 6 of stimula-tion in all treatment arms at a daily dose of 0.25 mg to prevent a premature LH surge. Suppression with the GnRH antagonist will be continued until the day of final oocyte maturation. Endocrine monitoring and ultrasound scan will be carried out on day 8 of stimulation and repeated every two days until trigger, de-pending on the patients' response. Triggering for final oocyte maturation is performed as soon as 3 follicles of ≥17 mm will be observed.

Cycles will be cancelled if less than 3 follicles of 12 mm are observed on day 8 day of stimulation, nonethe-less, blood test for hormonal evaluation will be performed in any case on day 8.

Oocyte maturation will be triggered with a single subcutaneous injection of hCG (Pregnyl®: 5000UI/sc, MSD, or 10000UI/sc if body weight exceeds 80 kg) as soon as 3 follicles of ≥17 mm will be observed. Ap-proximately 34-36 hours after trigger, oocyte retrieval will be performed. An embryo transfer will be per-formed on day 3 or on day 5 of embryonic development; one or 2 embryos will be replaced.

The luteal phase will be supported by vaginal administration of micronized progesterone 600 mg/day (Utrogestan®) from the day after ovarian puncture until the day of pregnancy test. In case of pregnancy, progesterone administration will be extended until week 7. In case of risk of OHSS, namely the presence of >18 follicles of 11 mm or more, final oocyte maturation will be triggered with a GnRH agonist (Gonapep-tyl, 0.2 mg) and a freeze-all strategy will be applied (Papanikolaou et al., 2006, Griesinger et al., 2016). A freeze -all strategy will also be applied in case of P>1.5 ng/mL on the day of hCG and per clinician prefer-ence.

All the patients will be asked to inject CFA and rFSH between 6-10 PM; the antagonist injection (ganirelix) will be performed between 7-11 AM and the endocrine profile measurements, alias blood tests, will be done between 7 and 11 AM.

ELIGIBILITY:
Inclusion Criteria

* Female age: > 18 to < 38 years
* The patient must have undergone not more than three consecutive unsuccessful IVF/ICSI cycles since the last ongoing pregnancy (whether fresh and/or several frozen ET resulted from these attempts)
* BMI ≤29 Kg /m2
* Patients of ≤ 35 years old, body weight should be ≥ 60kg
* Patients of >35 years old, body weight should be > 50 kg
* Regular normo-ovulatory menstrual cycles (26-35 days)
* Basal FSH <10 IU/l, basal E2 <60 pg/ml and basal Progesteone (< 1.5 ng/mL) (normal cycle day-3 basal serum hormone levels), to be measured on cycle day 2 or 3 of the treatment cycle
* Normal ultrasound scan (presence of both ovaries without evidence of abnormality within 6 months)
* AFC >7 and < 20
* No pill within the 3 months before treatment
* Signed informed consent

Exclusion Criteria

* Polycystic ovarian syndrome (PCOS) according to the Rotterdam classification (2004)
* Oocyte donors
* Poor responder patients (development of <4 follicles in previous IVF/ICSI or cancelled cycles)
* Endometriosis ≥ grade 3
* Contraindications to the use of gonadotropins
* Abnormal vaginal bleeding of unknown cause
* History of ovarian hyperstimulation syndrome (OHSS) or a previous ovarian stimulation cycle with more than 30 follicles of 11 mm or higher (as recommended by the Elonva® Summary of Product Characteristics)
* A history of recurrent miscarriage (three or more consecutive miscarriages)

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 261 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
serum progesterone level on the day of the trigger | 2 years
  Compare the mean serum progesterone level (ng/mL) on day of hCG between the study groups.

SECONDARY OUTCOMES:
Number of oocytes retrieved | 2 years
  number of oocytes retrieved the day of the pick up
Number of patients who underwent freeze all the embryos (FA) | 2 years
  number of patients who need to avoid the fresh embryo transfer (ET) and do a freeze all procedure.
Clinical pregnancy rate | 2 years
  The number of clinical pregnancies expressed per 100 initiated cycles, aspiration cycles or embryo transfer cycles. When clinical pregnancy rates are recorded, the denominator (initiated, aspirated or embryo transfer cycles) must be specified.
Miscarriage rate | 2 years
  Spontaneous loss of a clinical pregnancy before 22 completed weeks of gestational age, in which the embryo(s) or fetus(es) is/are nonviable and is/are not spontaneously absorbed or expelled from the uterus.

IPD SHARING:
Plan to Share IPD: No